CLINICAL TRIAL: NCT04620850
Title: Effect of Acupressure on Recovery of Bowel Function in Patients Post Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 165/2563
Record Dates: First submitted 2020-10-26; First posted 2020-11-09 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2020-09

CONDITIONS: Acupressure; Post-Op Complication; Cesarean Section; Bowel Ileus
MeSH Terms: conditions — Postoperative Complications; Ileus | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure (Experimental): Acupressure after cesarean section 3 hr and then next 3 hr (duration 10 min per time) Acupressure at below knee the point ai locate about4 finger spcae below patella on the lateral side of tibia bone
  Interventions: Device: Acupressure
- No acupressure (No Intervention): Standard post-operative care

INTERVENTIONS:
Device: Acupressure — Acupressure after cesarean section 3 hr and then next 3 hr (duration 10 min per time)
  Arms: Acupressure

SUMMARY:
Research objectives To compare the efficacy of acupressure with no acupressure to examine time to first flatus in patient post cesarean section

; Acupressure at ST-36 Zusanli (lateral to anterior crest of tibia, in the tibialis anterior muscle)

Research hypothesis Patients who received acupressure will have earlier flatus passage

DETAILED DESCRIPTION:
Research design Randomized controlled trial. Compare between The investigators is who assess the acupressure with control group is the participants do not assess the acupressure

ELIGIBILITY:
Inclusion Criteria:

1. Pregnancy woman age 18-45 years
2. General anesthesia
3. Co-operate in research
4. Can speak in thai language

Exclusion Criteria:

1. Twin pregnancy
2. Placenta previa
3. Placental abruption
4. Chorioamnionitis
5. Complication intraoperation (Bowel or bladder injury)
6. Post partum hemorrhage
7. Abdominal adhesion
8. Opertative time more than 2 hour
9. History gastrointestinal surgery
10. Prior acupressure
11. Neurological disease
12. Neuromuscular disease
13. Hepatic disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
To study the duration of the first time to flatus passage in post cesaren section patient | through study completion, an average of 1 year
  the duration ; hour after post cesaren section

SECONDARY OUTCOMES:
To study the duration of the first time to have bowel sound in post cesaren section patient | through study completion, an average of 1 year
  the duration ; hour after post cesaren section
To study the duration of the first time to pass stool in post cesaren section patient | through study completion, an average of 1 year
  the duration ; hour after post cesaren section
To study the symptomatic about Nausea/vomiting in post cesaren section patient | mild
  Score; mild,moderate,severe

CONTACTS AND LOCATIONS:
Overall Officials: Sasiwimol kunnitikorn, MD, Study Chair — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand